CLINICAL TRIAL: NCT02451956
Title: Study of AZD5363 in Combination With Paclitaxel, in Advanced Gastric Adenocarcinoma Patients Harboring PIK3CA Mutation and/or PIK3CA Amplification as a Second-line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-04-128
Record Dates: First submitted 2015-05-14; First posted 2015-05-22 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — capivasertib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD5363 in combination with paclitaxel (Experimental): AZD5363 400mg bid 4 days on/ 3 days off of a 7 day cycle for each week that paclitaxel is given + paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle. AZD5363 and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.If paclitaxel therapy is stopped then AZD5363 can be given on a 4on/3off continuous schedule.
  Interventions: Drug: AZD5363; Drug: paclitaxel

INTERVENTIONS:
Drug: AZD5363 — Dosage and Schedule : AZD5363 400mg bid 4 days on/ 3 days off of a 7 day cycle for each week
Drug: paclitaxel — paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle.

SUMMARY:
This study is a single arm, single center phase II study of AZD5363 in combination with paclitaxel in patients with advanced gastric adenocarcinoma harboring PIK3CA mutation or amplification as a second line chemotherapy.

Patients will receive AZD 5363 plus weekly paclitaxel combination regimen. A arm is composed of 25 patients.

Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date of enrollment, up to week 40, then every 16 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

Study treatment will be continued until objective disease progression.

DETAILED DESCRIPTION:
AZD5363 is a highly potent adenosine triphosphate (ATP)-competitive AKT inhibitor with IC50<10nmol/l for all three AKT isoforms.

AZD5363 is well designed to inhibit the important main signal pathway in various human cancer. AZD5363 is a specific inhibitor of the AKT pathway which is activated in a wide spectrum of tumours.The combination of AZD5363 to standard chemotherapy, paclitaxel, might improve the outcomes of 2nd line therapy in advanced gastric cancer patients .

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after first-line therapy.

   * The 1st line regimen must have contained doublet 5-fluoropyrimidine and platinum based regimen.
   * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doublet 5-fluoropyrimidine and platinum-based regimen could be considered as 1st line therapy.
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the 1st line therapy.
5. Provision of tumor sample (from either a resection or biopsy)
6. Patients with PIK3CA mutation and/or PIK3CA amplification
7. Eastern Cooperative Oncology Group performance status 0-1.
8. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
9. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥9.0 g/dL (transfusion allowed)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥100 x 109/L (transfusion allowed)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN
10. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
11. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1.

    Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.
12. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.

   * In case of investigator's discretion, patient has a specific biomarker and meets all eligible criteria except for line of therapy, patient will be allowed. However, only 3rd line is allowed in this isolated cases. In the case of other, PI should confirm.
2. Any previous treatment with PIK3CA and/or AKT inhibitors or agents with mixed PI3K / mTOR activity.
3. Any previous treatment with paclitaxel
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
5. HER2 positive patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)
6. Patients unable to swallow orally administered medication.
7. Any investigational drug or product administered within 30 days or 5 half-lives, whichever is longer, of the first dose of AZD5363.
8. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
9. Previous major surgery within 4weeks prior to first dose.
10. With the exception of alopecia, any ongoing toxicities (>Common Toxicity Criteria for Adverse Effects grade 1) caused by previous cancer therapy.
11. Intestinal obstruction or Common Toxicity Criteria for Adverse Effects grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
12. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
13. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Left ventricular ejection fraction <55% measured by echocardiography, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment.
14. Active or untreated brain metastases or spinal cord compression Patients with treated brain metastases or spinal cord compression are eligible if they have minimal neurologic symptoms, evidence of stable disease (for at least 1 month) or response on follow-up scan, and require no corticosteroid therapy for ≥ 1 week.
15. Patients with proteinuria (3+ on dipstick analysis )
16. Female patients who are breast-feeding or child-bearing
17. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
18. Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Object response rate (ORR) | expected average of 24 weeks

SECONDARY OUTCOMES:
Duration of response | expected average of 24 weeks
Disease control rate | 8 weeks
Overall survival | expected average of 24 weeks
progression-free survival | expected average of 24 weeks
Number of subjects with Adverse Events as a Measure of safety and tolerability | up to 100 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea